CLINICAL TRIAL: NCT03996551
Title: ExeRTiOn2- The Weight Gain Prevention Exercise in Renal Transplant Online Study. A Feasibility Randomised Controlled Trial.
Brief Title: ExeRTiOn2- The Weight Gain Prevention Exercise in Renal Transplant Online Study
Acronym: ExeRTiOn2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Kidney Research U.K. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KCH-ExeRTiOn2
Record Dates: First submitted 2019-06-18; First posted 2019-06-24 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Kidney Transplant; Complications; Weight Gain
Keywords: kidney transplant; weight gain prevention; behavior change techniques; dietary advice; physical activity advice
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will receive access to the 12-week kidney transplant specific weight gain prevention online resource (ExeRTiOn online resource). After the 12 weeks, they will be offered the option to continue using the website up until the completion of the study (12 months)
  Interventions: Behavioral: ExeRTiOn online resource
- Control group (No Intervention): This group will not receive the online resource. They will receive the standard encouragement to follow a healthy diet and perform physical activity during routine transplant follow up appointments.

INTERVENTIONS:
Behavioral: ExeRTiOn online resource — This is a 12-week online resource, specifically designed for new kidney transplant recipients. It includes dietary advice, physical activity advice, and recognized behavior change techniques. The participant will be monitored by a specialist physiotherapist and will receive messages of encouragement a 6 weeks and 12 weeks.
  Arms: Intervention Group

SUMMARY:
The primary aim of this trial is to assess the feasibility of a novel online weight gain prevention resource for new kidney transplant recipients at two London transplant clinics. A previous study conducted by the research team titled 'ExeRTiOn' provided usability feedback that led to revisions of this online resource in a purposive sample of kidney transplant recipients (n=11) and transplant multidisciplinary team members (n=6).

DETAILED DESCRIPTION:
This current study aims to recruit a sample of new kidney transplant recipients (n=50) from two transplant sites in London. Participants will be randomized to either the 12-week kidney transplant specific novel online weight gain prevention resource (n=25) or usual care (n=25). All participants will be assessed at baseline, 12 weeks and 12 months. The primary outcome of this study is feasibility (screening, recruitment, randomization, retention, adherence to the intervention and adherence to the study visits). The research team will also assess the ability to collect measures for a definitive study (body weight, body mass index, body composition, quality of life, self-efficacy, fatigue, arterial stiffness and physical function).

A nested qualitative study will capture participant experience at two time points during this 12 month trial. At 3 months semi-structured individual interviews will be conducted in a purposive approximately 6 to 10 of the intervention participants until data saturation is achieved. These interviews will assess the experience of using the online intervention. At 6 months a purposive sample of approximately 16 participants from both groups will complete individual semi-structured interviews to assess the experiences of participating in this trial.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or above
* able to provide written consent
* less than 3 months post kidney transplant
* access to the internet connected computer, tablet, laptop or smartphone
* a body mass index greater than or equal to 18.5 (healthy range)

Exclusion Criteria:

* age < 18
* current pregnancy
* unstable medication condition such as uncontrolled angina
* participation in a recent structured exercise programme in the last 3 months
* BMI of less than 18.5 (classified as underweight)
* significant cognitive impairment preventing them from engaging with the online resource
* unable to complete the resource in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility- screening of participants | through study completion, an average of 1 year
  number of participants screened per month, and those unwilling to take part
Feasibility- recruitment of participants into the trial | through study completion, an average of 1 year
  number of participants recruited per month
Feasibility- proportion of participants willing to be randomized | through study completion, an average of 1 year
  willingness of participants to be randomized to each group
feasibility- monthly retention of participants over the trial period | through study completion, an average of 1 year
  number of participants retained per month
feasibility- total retention of participants over the trial period | through study completion, an average of 1 year
  number of participants retained and at end of study
feasibility-adherence to ExeRTiOn online resource (intervention group) | by three months
  aim for 60% completion of sessions
feasibility- time taken to complete all study visits | through study completion, an average of 1 year
  the average time taken to complete study visits will be captured
feasibility- adherence to study visits throughout the trial | through study completion, an average of 1 year
  the proportion of completed study visits for outcome measures will be calculated
feasibility- safety throughout the trial | 12 months
  the number of hospital admissions (non-elective, or elective staying >24 hours) will be captured
feasibility- qualitative experience of participants using the online resource | 3 months
  individual semi-structured interviews in a purposive sample from the treatment group
feasibility- qualitative experience of participants participation in the trial | 6 months
  individual semi-structured interviews in a purposive sample of study participants

SECONDARY OUTCOMES:
change in body weight in kilograms over the trial | baseline, 3 months and 12 months
  body weight in kilograms will be recorded at the three study visits and the change will be calculated
body mass index over the 12 month trial | baseline, 3 months, 12 months
  body mass index at each 3 study visits
body composition over the 12 month trial | baseline, 3 months, 12 months
  body composition will be measured at each of the 3 study visits
quality of life (self-reported) over the 12 month trial | baseline, 3 months, 12 months
  QOL will be measured by the EQ5D questionnaire at each of the 3 study visits
self reported self-efficacy for nutrition scale over the 12 month trial | baseline, 3 months, 12 months
  self-efficacy for nutrition will be measured via the self-efficacy scale at each of the 3 study visits. The scale has 5 statements/questions. The user selects a number from 1 to 4, with 1 being very uncertain and 4 being very certain for each of the five statements. The highest score (higher self-efficacy) is 20, the lowest score (low self-efficacy) is 5.
self reported self-efficacy for physical exercise scale over the 12 month trial | baseline, 3 months, 12 months
  self-efficacy for physical exercise will be measured via this self-efficacy scale at each of the 3 study visits. The scale has 5 statements/questions. The user selects a number from 1 to 4, with 1 being very uncertain and 4 being very certain for each of the five statements. The highest score (higher self-efficacy) is 20, the lowest score (low self-efficacy) is 5.
Total score self reported fatigue via the Chalder Fatigue Questionnaire over the 12 months | baseline, 3 months, 12 months
  self-reported fatigue will be measured using the Chalder Fatigue scale. It has 11 items, 7 measure physical fatigue and 4 measure mental fatigue. The user rates each question on a likert scoring system 0-3, with the maximum score being 33 (high fatigue).
Physical fatigue (sub-scale) of the Chalder Fatigue Questionnaire over the 12 months | baseline, 3 months, 12 months
  7 of the items measure physical fatigue, the maximum sub score is 21(high physical fatigue)
Mental fatigue (sub-scale) of the Chalder Fatigue Questionnaire over the 12 months | baseline, 3 months, 12 months
  4 of the items measure mental fatigue, the maximum sub score is 12 (high mental fatigue)
arterial stiffness over the 12 month trial | at baseline, 3 months and 12 months
  arterial stiffness will be measured by pulse wave velocity
physical function over the 12 month trial | baseline, 3 months, 12 months
  physical function will be assessed by the six minute walk test at each timepoint

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Guy's and St Thomas' Hospital, London, UK
  - King's College Hospital, London, UK

IPD SHARING:
Plan to Share IPD: Undecided
The research team plans to publish the results in a journal publication. They will include anoymized raw data in the supplementary material

REFERENCES:
- [Derived] Castle EM, Dijk G, Asgari E, Shah S, Phillips R, Greenwood J, Bramham K, Chilcot J, Greenwood SA. The Feasibility and User-Experience of a Digital Health Intervention Designed to Prevent Weight Gain in New Kidney Transplant Recipients-The ExeRTiOn2 Trial. Front Nutr. 2022 May 23;9:887580. doi: 10.3389/fnut.2022.887580. eCollection 2022. PMID 35677553